CLINICAL TRIAL: NCT06872879
Title: The EFFECT of SIMULATION-BASED TRAINING with TWO DIFFERENT REALITY LEVELS on POSTPARTUM HAEMORRHAGE MANAGEMENT SKILLS in NURSING STUDENTS
Brief Title: The EFFECT of SIMULATION-BASED TRAINING on POSTPARTUM HAEMORRHAGE MANAGEMENT SKILLS
Acronym: (SBT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Yılda Arzu Aba, Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-128
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Simulation Training; Nursing; Postpartum Hemorrhage
Keywords: Simulation Training; Nursing; Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: The study was a parallel design randomised comparative study designed with equality experiment to determine the effect of simulation-based training using two different reality levels (visually enhanced mental simulation (VEMS) and hybrid simulation) on PPH management skills in nursing students.
Who Masked: Outcomes Assessor
Masking Description: Since the researcher is implementing the educational interventions and the students are aware of the interventions in the study, blinding will not be performed in this study. However, during the data analysis phase, the groups will be named as 1 and 2. Thus, the researcher performing the data analysis will be blinded to the type of intervention applied to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Students in the VEMS (Visually Enhanced Mental Simulation) group will receive a structured training programme to improve their PPH management skills.
  Interventions: Other: VEMS Simulation
- Group 2 (Active Comparator): Students in the hybrid simulation group will receive a simulation-based training in which the standard patient and part task trainer are used together.
  Interventions: Other: Hybrit Simulation

INTERVENTIONS:
Other: VEMS Simulation — Students in the VEMS (Visually Enhanced Mental Simulation) group will receive a structured training programme to improve their PPH management skills. This process consists of three main stages: Theoretical training, skills training and simulation practice.
  1.1 hour theoretical training will be given to the students to remind them the basic information about PPH management.
  2. PPH management will be mentally visualised step by step using VEMS materials. Students will be individually involved in the scenario and will apply the steps of PPH management in a mental simulation environment. After the scenario is completed, a 30-minute debriefing session will be organised.
  3. Manikin simulation will be used to evaluate students' PPH management skills. Students' PPH management skills will be evaluated using the "Postpartum Haemorrhage Management Observation Form". Attitudes towards the learning process will be measured by applying the Student Satisfaction and Confidence in Learning Scale.
  Arms: Group 1
Other: Hybrit Simulation — Students in the hybrid simulation group will receive a simulation-based training in which the standard patient and part task trainer are used together. This process consists of three main stages: theoretical training, skills training and simulation practice.
  1.1 hour theoretical training to remind basic information about PPH management. 2. Standard patient and part task trainers will be used in the skills training of the students. Students will make patient assessment, check vital signs and plan necessary interventions by contacting the standard patient.After the scenario is completed, a 30-minute debriefing session will be organised.
  3. Manikin simulation will be used to evaluate students' PPH management skills. Students' PPH management skills will be evaluated using the "Postpartum Haemorrhage Management Observation Form". Attitudes towards the learning process will be measured by applying the Student Satisfaction and Confidence in Learning Scale.
  Arms: Group 2

SUMMARY:
This study was planned to determine the effect of simulation-based training using two different reality levels-visually enhanced mental simulation (VEMS) and hybrid simulation-on postpartum haemorrhage (PPH) management skills in nursing students.

DETAILED DESCRIPTION:
This study will be conducted to determine the effect of simulation-based training using two different reality levels-visually enhanced mental simulation (VEMS) and hybrid simulation-on postpartum haemorrhage (PPH) management skills in nursing students. PPH is one of the leading causes of postpartum maternal mortality and its effective management requires the knowledge, skills and coordination of the healthcare team. However, it is difficult for nursing students to acquire these skills directly in the clinical environment due to rare observation and structural limitations in education. Simulation-based education stands out as an important method to develop such critical clinical skills.

In this randomised comparative study, 4th year students studying at Bandırma Onyedi Eylül University, Department of Nursing who have completed the course of Women's Health and Diseases Nursing in the spring semester of the 2024-2025 academic year will be included in the study. The sample size was calculated by G*Power analysis and a total of 64 students were randomly assigned to two groups. One of the intervention groups will receive PPH management training with VEMS method and the other will receive PPH management training with hybrid simulation. The training programme will be conducted within the scope of a structured curriculum including theoretical training, skills training and simulation applications.

'Participant Information Form', "Postpartum Haemorrhage Management Observation Form" and "Student Satisfaction and Confidence in Learning Scale" will be used to collect data. The skill levels of the students will be evaluated by two independent observers, and learning satisfaction and self-confidence levels will be measured through the scales.

The findings of the study are expected to provide important contributions in evaluating the effect of simulation-based training on PPH management skills. In particular, it is investigated whether the low-cost and highly applicable VEMS method is effective in terms of student satisfaction, confidence in learning and skill development as an alternative to traditional simulation approaches. The results obtained from the study may provide evidence-based recommendations to increase the efficiency of simulation applications in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* To have a grade point average of 2.00 and above

Exclusion Criteria:

* Not participating in all stages of the training programme
* Incomplete completion of data collection tools
* Wanting to leave the research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
PPH management skill levels | 2 weeks after the completion of the simulation training
  The form, which enables the assessment of students' skills in the PPH management process, consists of 25 steps.
Satisfaction and self-confidence levels in learning | 2 weeks after the completion of the simulation training
  Student Satisfaction and Confidence in Learning Scale will be used.

IPD SHARING:
Plan to Share IPD: No